CLINICAL TRIAL: NCT07046910
Title: Advanced Immunoclinical Phenotyping of Rejection in Lung Transplant
Brief Title: Developing Hyperpolarized Gas MRI Signatures to Detect and Manage Acute Cellular Rejection
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Y. Michael Shim, MD, Professor of Pulmonary and Critical Care Medicine, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20987-3; R01HL173369-01 (NIH)
Record Dates: First submitted 2025-06-14; First posted 2025-07-02 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Lung Transplant Rejection
Keywords: lung transplant; hyperpolarized xenon-129 MRI; bronchoscopy

STUDY DESIGN:
Intervention Model Description: Part 3 Substudy: Testing the diagnostic performance of tissue pathology from blood, urine, and BAL from clinical bronchoscopy with vs. without hyperpolarized Xenon MRI. Determining the HXe MRI responses between before and after ACR treatment. Testing the correlation between HGMRI and scRNA-sequence from areas with vs. without ACR.Testing the correlation between HGMRI and scRNA-sequence and testing the agreement between the diagnoses by HXe MRI vs. tissue pathology from clinical navigational bronchoscopy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Substudy(Active): Two Longitudinal Lung MRI study with two navigational Bronchoscopy (Experimental): * blood
  * urine
  * Two navigational bronchoscopies and two MRIs for tissue
  Interventions: Diagnostic Test: Sub study (Active): Two Lung MRI study with two navigational Bronchoscopy; Drug: Hyperpolarized Xenon129

INTERVENTIONS:
Diagnostic Test: Sub study (Active): Two Lung MRI study with two navigational Bronchoscopy — Hyperpolarized Xenon-129 MRI twice with navigational bronchoscopy twice
  Other Names: Lung transplant recipient without HXe MRI prior to navigational bronchoscopy
Drug: Hyperpolarized Xenon129 — Lung transplant recipient with hyperpolarized Xe129 in MRI as an inhalation contrast agent
  Other Names: MRI

SUMMARY:
Lung transplantation (LT) is the only definitive therapy for many patients with end-stage lung diseases. The supply of donors' lungs is the biggest bottleneck to performing a lung transplant, and many patients die while waiting. Acute Cellular Rejection (ACR) is a significant risk factor for developing chronic allograft failure, a primary reason for death in this patient population. These observations highlight the importance of early diagnosis and management of ACR to prevent chronic graft failure. The preliminary results support the idea that Hyperpolarized Gas Magnetic Resonance Imaging has excellent potential to address this clinical gap. This study hypothesizes that optimized hyperpolarized gas magnetic resonance imaging (HGMRI) signatures can detect early pathophysiologic derangements in lung allografts consistent with ACR. This study also hypothesizes that the optimized HGMRI signatures will correlate with single-cell transcriptomic signatures that reflect dysregulated immune responses associated with ACR.

DETAILED DESCRIPTION:
Lung transplantation (LT) is the only definitive therapy for subjects with end-stage lung diseases. The supply of donors' lungs is the biggest bottleneck to performing a lung transplant, and many patients die while waiting. Many lung transplant recipients experience at least one acute rejection episode after transplantation. Acute Cellular Rejection (ACR) is a significant risk factor for developing chronic allograft failure, a primary reason for death in this patient population. These observations highlight the importance of early diagnosis and management of ACR to prevent chronic graft failure. The preliminary results support the idea that Hyperpolarized Gas Magnetic Resonance Imaging (HGMRI) signatures have excellent potential to address this clinical gap. In lung transplant patients without suspicion of ACR, HGMRI detected subtle, regional abnormalities in pulmonary physiology that were not detected by pulmonary function tests (PFTs) or high-resolution chest computer tomography (HRCT). Biopsy-proven regions of ACR in these subjects exhibited worse airflow and gas exchange HGMRI signatures, which corroborated well with the tissue pathology diagnosis of ACR. This data demonstrates the potential of HGMRI signatures to detect ACR even when existing clinical tools cannot. By merging anatomic CT and physiologic HGMRI readouts, the previous study developed a method to identify the airways that led to the allograft segments with abnormal HGMRI signatures. Then, a method to sample these areas of allografts is enabled during routine surveillance bronchoscopy by mapping the airways leading to dysfunctional allograft regions to enhance the diagnostic accuracy of clinical bronchoscopy. The primary molecular driver of ACR is the exaggerated host immune response to the donor's lungs. The anticipated results are that within the same subject, the single-cell transcriptome of cells from lung regions with abnormal HGMRI signatures would be more immunologically abnormal than those with normal HGMRI signatures. The hypothesis is that optimized HGMRI signatures can detect early pathophysiologic derangements in lung allografts consistent with ACR. The second hypothesis is that the optimized HGMRI signatures correlate with single-cell transcriptomic signatures reflecting the dysregulated immune responses underlying ACR. This study proposes: Aim 1: Determine the optimized HGMRI signatures to detect early regional allograft dysfunction consistent with ACR in lung allografts at the baseline Visit 1 (V1); Aim 2: Determine how the within-subject longitudinal changes in regional HGMRI signatures over a 1-year follow-up Visit 2 (V2) correlate with a clinical diagnosis of ACR.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be willing to participate and undergo the procedure, and be managed as outpatients
* HXe MRI-specific Inclusion
* All patients who successfully underwent a lung transplant at the University of Virginia
* Followed by the medical lung transplant team for the post-lung transplant rejection surveillance program at the University of Virginia
* a clinical diagnosis of lung transplant within the past 12 months
* absence of any significant allograft dysfunction/rejection at the time of the 12-month surveillance bronchoscopy
* the ability to understand a written informed consent form and comply with the requirements of the study.
* have an acceptable pre-bronchoscopy pulmonary function test: FEV1>45% before use of any bronchodilator
* Must have acceptable pre-procedural screening studies.
* Complete Blood Count: normal WBC, Hgb, and PLT
* PT: Normal < 1.2
* Basic Metabolic Panel: Normal

  1. Scenario 1 (two visits): Standard bronchoscopy with Normal MRI results and without a diagnosis of acute rejection after bronchoscopy.
  2. Scenario 2 (two visits): Navigational bronchoscopy with abnormal MRI result but without a diagnosis of acute rejection after bronchoscopy by clinical pathology.
  3. Scenario 3 (three or four visits): Navigational bronchoscopy with abnormal MRI result and a diagnosis of acute rejection after bronchoscopy by clinical pathology at the first visit, the second visit, or both visits.
  4. Scenario 4 (one visit): Subjects who previously signed Part 2 Substudy corresponding to the First HXe MRI visit of the Part 3 Substudy (6 or 12 month evaluation). They will be asked to join the Part 3 Substudy to undergo a 24-month follow-up evaluation, including MRI and bronchoscopy, as described for Scenarios 1, 2, or 3.

     Exclusion Criteria:

  <!-- -->

  1. Unable to Consent
  2. Continuous oxygen use at home.
  3. Blood oxygen saturation of less than 92% as measured by pulse oximetry on the day of imaging.
  4. FEV1 percent predicted less than 25%.
  5. Pregnancy or lactation.
  6. Claustrophobia, inner ear implants, aneurysms or other surgical clips, metal foreign bodies in the eye, pacemakers, or other contraindications to MR scanning. Subjects with any implanted device that cannot be verified as MRI compliant will be excluded.
  7. Chest circumference greater than that of the xenon MR and/or helium coil. The circumference of the coil is approximately 42 inches.
  8. History of congenital cardiac disease, chronic renal failure, or cirrhosis.
  9. Inability to understand simple instructions or to hold still for approximately 10 seconds.
  10. History of respiratory infection within 2 weeks prior to the MR scan
  11. History of MI, stroke, and/or poorly controlled hypertension.
  12. Failure to complete study-related procedures
  13. Unavailability of a reliable communication network and contacts for follow-up with the second in-house backup contact
  14. Patient actively smokes.
  15. Before 48 hours, any event being considered to be too risky to preclude surveillance bronchoscopy: SaO2 <90%, >16 puffs/24 hours of short-acting β-agonist (SABA), worsening symptoms prompting the use of any inhalers, FEV1 < 45% before using a bronchodilator.
  16. acute or chronic renal failure
  17. uncontrolled coronary artery disease or congestive heart failure; uncontrolled diabetes mellitus; uncontrolled hypertension, liver disease; history of neurologic diseases, including stroke, any disease concerning fibrotic processes.
  18. Pregnant females will be excluded
  19. Claustrophobic or too large to fit into the available MR chest RF coils.

      -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of Ventilation Defect Percent by MRI (continuous variable %VDP) | 6 or 12 months then 24 months after the date of lung transplant surgery
  The outcome of Airway abnormalities suggestive of acute rejection
Measurement of Lung gas exchange capacity by MRI (continuous variable of red blood cell gas exchange function called RBC/Gas) | 6 or 12 months then 24 months after the date of lung transplant surgery
  The outcome of Lung parenchymal gas exchange abnormalities suggestive of acute rejection
Measurement of the Single-cell RNA-sequencing of the bronchoalveolar lavage cells (Top 25 gene signatures over-expressed in lung area with acute rejection) | 6 or 12 months then 24 months after the date of last HXe MRI
  What the Single-cell transcriptomic signatures being suggestive of acute rejection
Measurement of Pulmonary function test (Spirometry) | 6 or 12 months then 24 months after the date of last HXe MRI
  Determining what the Clinical pulmonary function test suggestive of acute rejection

CONTACTS AND LOCATIONS:
Overall Officials: Yun M Shim, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual-level data will be made available at publication or at the time of study completion per the funding agency's policy (NIH/NHLBI).
Supporting Information: CSR
Time Frame: Either at the time of data publication or after the study completion.
Access Criteria: The access request must meet minimal criteria, such as being a qualified researcher with an approved data-sharing agreement with a research analysis plan. The basic policy is referred to NIH data-sharing policy (funding agency)
URL: https://sharing.nih.gov/data-management-and-sharing-policy/about-data-management-and-sharing-policies/data-management-and-sharing-policy-overview#after